CLINICAL TRIAL: NCT03772834
Title: A Combination Therapy to Treat Cancer-Related Fatigue - NCI R01
Brief Title: Methylphenidate and Exercise in Reducing Cancer-Related Fatigue in Patients With Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018-0559; NCI-2018-02527 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0559 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group I (methylphenidate, resistance training, walking) (Experimental): Patients receive methylphenidate PO BID and undergo exercise program consisting of resistance training BIW and walking 15- 40 minutes a day 4 days a week for 12 weeks.
  Interventions: Behavioral: Exercise Intervention; Drug: Methylphenidate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (placebo, resistance training, stretching) (Active Comparator): Patients receive a placebo PO BID and undergo exercise program consisting of resistance training BIW and walking 15-40 minutes a day for 4 days a week for 12 weeks.
  Interventions: Behavioral: Exercise Intervention; Other: Placebo; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group III (methylphenidate, stretching) (Active Comparator): Patients receive methylphenidate PO BID and undergo stretching for 4 days a week for 12 weeks.
  Interventions: Drug: Methylphenidate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Stretching
- Group IV (placebo, stretching) (Active Comparator): Patients receive a placebo PO BID and undergo stretching for 4 days a week for 12 weeks.
  Interventions: Other: Placebo; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Stretching

INTERVENTIONS:
Behavioral: Exercise Intervention — Undergo resistance training and walking
  Arms: Group I (methylphenidate, resistance training, walking); Group II (placebo, resistance training, stretching)
Drug: Methylphenidate — Given PO
  Other Names: Daytrana
  Arms: Group I (methylphenidate, resistance training, walking); Group III (methylphenidate, stretching)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Group II (placebo, resistance training, stretching); Group IV (placebo, stretching)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Stretching — Undergo stretching
  Arms: Group III (methylphenidate, stretching); Group IV (placebo, stretching)

SUMMARY:
This phase II/III trial studies how well methylphenidate and exercise work in reducing cancer-related fatigue in patients with prostate cancer. Methylphenidate is a type of central nervous system stimulant that can improve cognitive ability, mainly in memory and cognitive function. Exercise can improve mood and the physical aspects of cancer-related fatigue. Giving methylphenidate in combination with exercise may work better in reducing cancer-related fatigue in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the combination of exercise (EX) plus methylphenidate (MP) is superior to exercise plus placebo in the treatment of cancer-related fatigue (CRF) in patients with prostate cancer scheduled to receive radiotherapy with androgen deprivation therapy for 12 weeks.

SECONDARY OBJECTIVE:

I. To determine the effects of combined exercise plus methylphenidate on quality-of-life, mood, physical, and cognitive measures.

EXPLORATORY OBJECTIVES:

I. To identify potential synergistic effects of exercise and methylphenidate in improvement of CRF.

II. To explore changes in brain activity by electroencephalography (EEG) in responders (with 4 point or greater change in Functional Assessment of Chronic Illness Therapy-Fatigue [FACIT-F] scores) versus (vs) non-responders to the intervention.

OUTLINE: Patients are randomized to 1 of 4 groups.

GROUP I: Patients receive methylphenidate orally (PO) twice daily (BID) and undergo exercise program consisting of resistance training twice weekly (BIW) and walking 15- 40 minutes a day 4 days a week for 12 weeks.

GROUP II: Patients receive a placebo PO BID and undergo exercise program consisting of resistance training BIW and walking 15-40 minutes a day for 4 days a week for 12 weeks.

GROUP III: Patients receive methylphenidate PO BID and undergo stretching for 4 days a week for 12 weeks.

GROUP IV: Patients receive a placebo PO BID and undergo stretching for 4 days a week for 12 weeks.

After completion of study treatment, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of prostate cancer and be scheduled to receive radiotherapy with concurrent androgen deprivation therapy, and presence of fatigue with severity of 1/10, on a 0-10 scale for at least 2 weeks
* Patient not regularly engaging in moderate aerobic exercise for >90 minutes/week and/or vigorous aerobic exercise for >30 minutes/week, and/ or strength training for >/= 1 day/week
* Have no clinical evidence of cognitive failure as evidenced by Memorial Delirium Assessment Scale score of </=13 at baseline
* Be aged 18 years or older
* Be willing to engage in follow-up telephone calls with a research staff
* Be willing to participate in the exercise programs
* Have telephone access so they can be contacted by the research staff
* Have a hemoglobin level of >/= 10 g/dL within 2 weeks of enrollment
* Be able to understand the description of the study and give written informed consent
* Have a Zubrod performance status score of 0 to 2
* Seen at an outpatient clinic at MD Anderson Cancer Center, its Houston Area Locations (HALs) or Smith Radiation Oncology Clinic (HHS)

Exclusion Criteria:

* Have a major contraindication to MethylphenidateMP) (e.g., allergy/hypersensitivity to study medications or their constituents), exercise (e.g., cardiac disease), or conditions making adherence difficult as determined by the attending physician
* Be currently taking MP, or have taken it within the previous 10 days
* Be unable to complete the baseline assessment forms (e.g., due to language or sensory barriers) or to understand the recommendations for participation in the study
* Need monoamine oxidase inhibitors, tricyclic antidepressants, or clonidine
* Have glaucoma
* Have severe cardiac disease (New York Heart Association functional class III or IV)
* Have tachycardia and/or uncontrolled hypertension
* Be currently receiving anticoagulants, anticonvulsants (phenobarbital, diphenylhydantone, primidone), phenylbutazone, and/or tricyclic drugs (imipramine, clomipramine, or desipramine).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Level of cancer-related fatigue in all groups | Up to 12 weeks
  Will measure cancer-related fatigue (CRF) using the area under the curve (AUC) of the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) subscale score. The intervention exposure will be operationalized as proportion of the total minutes of prescribed exercise intervention the study patient was actually able to participate, or the proportion of prescribed study medication the study patient was able to actually take.

SECONDARY OUTCOMES:
Change in quality of life, mood, physical and cognitive measures in all groups | Baseline up to 12 weeks
  Will use a mixed-effects model to compare changes in Functional Assessment of Cancer Therapy - General (FACT-G), Pittsburgh Sleep Quality Index (PSQI), Multidimensional Fatigue Symptom Inventory - Short Form (MFSI-SF), Hospital Anxiety and Depression Scale (HADS), usual gait speed, hand grip strength (HGS), 30 second chair stand test (30s-CST), actigraphy, VO2 max, and C-reactive protein scores over time between the four treatment groups. For the mixed effects model, we will estimate the slopes for the changes in scores over time for each group and test the difference in these slopes.

OTHER OUTCOMES:
Synergistic effects of methylphenidate and exercise in all groups | Up to 12 weeks
  Will measure the synergistic effects of methylphenidate and exercise in improving CRF using the AUC of the FACIT-F subscale score. The analysis will be conducted using a linear model with the AUC as the response variable and indicator variables for the exercise and methylphenidate main effects as well as a product term of these indicator variables to assess the magnitude of synergy.
Change in brain activity by electroencephalography (EEG) in responders versus non-responders as measured by the FACIT-F score | Baseline up to 12 weeks
  Responders are identified as those who report a 4 point or greater change, while non-responders report less than a 4 point change in the FACIT-F score. EEG data will be grouped according to response status. Between-group differences will be examined using univariate analysis of variance (ANOVA) with condition (responders or non-responders) as the fixed factor of interest, and the change of power from baseline to the resting state EEG at day 29 and day 84 as the dependent variable. Additional analyses will include analysis of covariance (ANCOVA) by adjusting for baseline covariates including age, stage of disease, total dose of radiotherapy, and other covariates as necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org